CLINICAL TRIAL: NCT04178941
Title: Feasibility Pilot of Audit and Feedback With Educational Outreach to Align Continuous Pulse Oximetry Use in Stable Bronchiolitis With Evidence and Guideline Recommendations
Brief Title: Aligning Pulse Oximetry With Guidelines
Acronym: EMO Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-016718; 5U01HL143475-02 (NIH)
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Single Arm) (Experimental): The intervention is a combined educational outreach and audit and feedback strategy that includes providing the hospital's own continuous pulse oximetry use data back to them on a weekly basis. The data will be accompanied by staff-targeted educational materials and outreach sessions summarizing the current evidence and guideline recommendations for continuous pulse oximetry use in bronchiolitis.
  Interventions: Behavioral: Audit and Feedback; Behavioral: Educational outreach

INTERVENTIONS:
Behavioral: Audit and Feedback — The audit and feedback intervention includes providing each hospital's own continuous pulse oximetry use data back to them on a weekly basis for review and action.
Behavioral: Educational outreach — Educational outreach includes staff-targeted educational materials and outreach sessions summarizing the current evidence and guideline recommendations for continuous pulse oximetry use in bronchiolitis.

SUMMARY:
The primary objective is to measure the feasibility, acceptability, and appropriateness of audit and feedback with educational outreach as a strategy to align continuous pulse oximetry use in stable bronchiolitis patients with evidence and guideline recommendations.

DETAILED DESCRIPTION:
Continuous pulse oximetry (SpO2) monitoring has revolutionized detection of oxygen desaturation in operating rooms and other high-risk areas, improving outcomes in those settings. However, research suggests that overuse of continuous SpO2 monitoring in stable children with bronchiolitis who are unlikely to benefit from it is low-value care that places some children at risk of adverse outcomes. Despite national guidelines discouraging continuous pulse oximetry use in stable bronchiolitis patients, 46% of those infants and children are continuously monitored. This pragmatic, prospective, non-randomized, single-arm feasibility pilot will be performed on non-Intensive Care Unit (ICU) hospital units that care for bronchiolitis patients. The primary subjects are hospital staff who order or manage continuous pulse oximetry monitoring for bronchiolitis patients; secondary subjects are patients age 2 through 23 months with a primary diagnosis of bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Primary subjects - Hospital staff

  1. Nurses, physicians, physician assistants, nursing assistants, or respiratory therapists
  2. Providing care to patients on units included in the study.
* Secondary subjects - Patients

  1. Males or females 8 weeks through 23 months old hospitalized on non-Intensive Care Unit (ICU) wards
  2. Cared for by generalist inpatient services (e.g. general pediatrics, hospital medicine)
  3. Primary diagnosis of acute bronchiolitis according to hospital chart
  4. Not currently requiring supplemental oxygen therapy or nasal cannula flow at an fraction of inspired oxygen in the air (FiO2) of 21% (room air flow)

Exclusion Criteria:

* Primary subjects - Hospital staff

  1) None. Staff may self-exclude by choosing not to interact with the electronic communications and may choose to not attend meetings where the intervention is discussed.
* Secondary subjects - Patients

  1. Premature birth: <28 weeks completed gestation
  2. Cyanotic congenital heart disease
  3. Pulmonary hypertension
  4. Home oxygen or positive pressure ventilation requirement
  5. Tracheostomy
  6. Neuromuscular disease
  7. Immunodeficiency
  8. Cancer
  9. Historical, current, or suspected diagnosis of heart failure, myocarditis, or arrhythmia
  10. Historical, current, or suspected diagnosis of Coronavirus disease 2019 (COVID-19)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1898 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Bonafide, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faerber JA, Xiao R, Makeneni S, Schisterman EF, Brady PW, Schondelmeyer AC, Landrigan CP, Lucey K, Lee V, Gregory PF, Prasto J, Parthasarathy P, Greenfield M, Solomon C, Brent CR, Albanowski K, Beidas RS, Bonafide CP; Pediatric Research in Inpatient Settings (PRIS) Network. Sustainment of continuous pulse oximetry deimplementation: Analysis of Eliminating Monitor Overuse study data from six hospitals. J Hosp Med. 2023 Aug;18(8):724-729. doi: 10.1002/jhm.13154. Epub 2023 Jun 28. PMID 37380625
- [Derived] Schondelmeyer AC, Bettencourt AP, Xiao R, Beidas RS, Wolk CB, Landrigan CP, Brady PW, Brent CR, Parthasarathy P, Kern-Goldberger AS, Sergay N, Lee V, Russell CJ, Prasto J, Zaman S, McQuistion K, Lucey K, Solomon C, Garcia M, Bonafide CP; Pediatric Research in Inpatient Settings (PRIS) Network. Evaluation of an Educational Outreach and Audit and Feedback Program to Reduce Continuous Pulse Oximetry Use in Hospitalized Infants With Stable Bronchiolitis: A Nonrandomized Clinical Trial. JAMA Netw Open. 2021 Sep 1;4(9):e2122826. doi: 10.1001/jamanetworkopen.2021.22826. PMID 34473258

RESULTS

PARTICIPANT FLOW:
Groups:
- PATIENTS OBSERVED - Intervention (Single Arm): This arm refers to patients who were exposed to the intervention described below and who had their clinical data collected prospectively during the trial.
  The intervention is a combined educational outreach and audit and feedback strategy that includes providing the hospital's own continuous pulse oximetry use data back to them on a weekly basis. The data will be accompanied by staff-targeted educational materials and outreach sessions summarizing the current evidence and guideline recommendations for continuous pulse oximetry use in bronchiolitis.
  Audit and Feedback: The audit and feedback intervention includes providing each hospital's own continuous pulse oximetry use data back to them on a weekly basis for review and action.
  Educational outreach: Educational outreach includes staff-targeted educational materials and outreach sessions summarizing the current evidence and guideline recommendations for continuous pulse oximetry use in bronchiolitis.
- STAFF SURVEYED - Intervention (Single Arm): This arm refers to staff who were exposed to the intervention described below and who responded to the surveys administered for the feasibility, acceptability, and appropriateness outcome measures.
  The intervention is a combined educational outreach and audit and feedback strategy that includes providing the hospital's own continuous pulse oximetry use data back to them on a weekly basis. The data will be accompanied by staff-targeted educational materials and outreach sessions summarizing the current evidence and guideline recommendations for continuous pulse oximetry use in bronchiolitis.
  Audit and Feedback: The audit and feedback intervention includes providing each hospital's own continuous pulse oximetry use data back to them on a weekly basis for review and action.
  Educational outreach: Educational outreach includes staff-targeted educational materials and outreach sessions summarizing the current evidence and guideline recommendations for continuous pulse oximetry use in bronchiolitis.
Period: Overall Study
Arm/Group | PATIENTS OBSERVED - Intervention (Single Arm) | STAFF SURVEYED - Intervention (Single Arm)
Started | 1051 | 847
Completed | 1051 | 847
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: For the patients observed, 1051 matches the participant flow. For the staff surveyed, we include 847 which is the total number of surveys received and analyzed for the outcome measures specified.
Groups:
- Total: Total of all reporting groups
Arm/Group | PATIENTS OBSERVED - Intervention (Single Arm) | STAFF SURVEYED - Intervention (Single Arm) | Total
Number analyzed (Participants) | 1051 | 847 | 1898
Age, Customized [Count of Participants; unit: Participants]
  Age category: 8 weeks - 5 months old | 534 | 0 | 534
  Age category: 6 months - 11 months old | 284 | 0 | 284
  Age category: 12 months - 17 months old | 153 | 0 | 153
  Age category: 18 months - 23 months old | 80 | 0 | 80
  Age category: Unknown age | 0 | 847 | 847
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1049/1051 patients had sex data available in the medical record 818/847 survey respondents chose to disclose their sex
  Participants
    number analyzed (Participants) | 1049 | 818 | 1867
    Female | 438 | 695 | 1133
    Male | 611 | 123 | 734
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 305 | 77 | 382
  Not Hispanic or Latino | 609 | 703 | 1312
  Unknown or Not Reported | 137 | 67 | 204
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 38 | 161 | 199
  Native Hawaiian or Other Pacific Islander | 5 | 9 | 14
  Black or African American | 236 | 26 | 262
  White | 354 | 515 | 869
  More than one race | 15 | 30 | 45
  Unknown or Not Reported | 402 | 102 | 504

OUTCOME MEASURES:

1. Primary Outcome: Audit & Feedback Feasibility Using Adapted Item From Feasibility of Intervention Measure (FIM)
Description: The participant rates the feasibility of the intervention based on this statement: "Data feedback about our use of continuous pulse oximetry in patients with bronchiolitis is easy to implement." Data was only collected from the "STAFF SURVEYED - Intervention (Single Arm)" Arm/Group for this Outcome Measure.
Time Frame: 1 month after intervention
Population: 659 of the 847 overall respondents to the survey responded to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | STAFF SURVEYED - Intervention (Single Arm)
Number analyzed (Participants) | 659
Participants
  Completely agree | 222
  Agree | 331
  Neither agree nor disagree | 86
  Disagree | 20
  Completely diagree | 0

2. Primary Outcome: Audit & Feedback Acceptability Using Adapted Item From Acceptability of Intervention Measure (FIM)
Description: The participant rates the acceptability of the intervention based on this statement: "I like the data feedback." Data was only collected from the "STAFF SURVEYED - Intervention (Single Arm)" Arm/Group for this Outcome Measure.
Time Frame: 1 month after intervention
Population: 659/847 survey respondents answered this question.
Measure: Count of Participants; unit: Participants
Arm/Group | STAFF SURVEYED - Intervention (Single Arm)
Number analyzed (Participants) | 659
Participants
  Completely agree | 305
  Agree | 305
  Neither agree nor disagree | 46
  Disagree | 2
  Completely disagree | 1

3. Primary Outcome: Audit & Feedback Appropriateness Using Adapted Item From Intervention Appropriateness Measure (IAM)
Description: The participant rates the appropriateness of the intervention based on this statement: "Data feedback about our use of continuous pulse oximetry in bronchiolitis seems like a good match for our non-ICU floors that care for bronchiolitis." Data was only collected from the "STAFF SURVEYED - Intervention (Single Arm)" Arm/Group for this Outcome Measure.
Time Frame: 1 month after intervention
Population: 659/847 survey respondents answered this question.
Measure: Count of Participants; unit: Participants
Arm/Group | STAFF SURVEYED - Intervention (Single Arm)
Number analyzed (Participants) | 659
Participants
  Completely agree | 280
  Agree | 337
  Neither agree nor disagree | 37
  Disagree | 4
  Completely disagree | 1

4. Secondary Outcome: Hospital-level Percentage of Patients Continuously Monitored When Not Receiving Supplemental Oxygen
Description: Continuous pulse oximetry use rates in children with bronchiolitis who are not requiring supplemental oxygen administration. This is calculated as the number of patients continuously monitored when not receiving supplemental oxygen divided by the total number of patients observed when not receiving supplemental oxygen.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | PATIENTS OBSERVED - Intervention (Single Arm)
Number analyzed (Participants) | 1051
Participants | 236

5. Secondary Outcome: Sensitivity of the Presence of Electronic Health Record (EHR) Data From the Medical Monitoring Device for Actual Monitoring at the Bedside in Bronchiolitis. Sensitivity is Also Referred to as the "True Positive Rate."
Description: This measure will be calculated using chart review (to determine presence of electronic health record data from the medical monitoring device) and direct observation (to determine actual monitoring at the bedside). This outcome compared EHR data at minute 0 (same minute as direct observation occurred). The numerator is the number of patients with EHR data from the medical monitoring device.
  The denominator is the number of patients who were truly monitored.
Time Frame: 4 months
Population: The denominator of sensitivity is those patients who were truly monitored, which for this analysis was 102.
Measure: Count of Participants; unit: Participants
Arm/Group | PATIENTS OBSERVED - Intervention (Single Arm)
Number analyzed (Participants) | 102
Participants | 92

6. Secondary Outcome: Specificity of the Absence of Electronic Health Record Data From the Medical Monitoring Device for Absence of Monitoring at the Bedside in Bronchiolitis. Specificity is Also Referred to as the "True Negative Rate."
Description: This measure will be calculated using chart review (to determine presence of electronic health record data from the medical monitoring device) and direct observation (to determine actual monitoring at the bedside). This outcome compared EHR data at minute 0 (same minute as direct observation occurred). The numerator is the number of patients with absence of EHR data from the medical monitoring device. The denominator is the number of patients who were truly not monitored.
Time Frame: 4 months
Population: The denominator for specificity in this analysis was the number of patients who were truly not monitored, which was 566 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | PATIENTS OBSERVED - Intervention (Single Arm)
Number analyzed (Participants) | 566
Participants | 554

7. Secondary Outcome: Positive Predictive Value (PPV) of the Presence of Electronic Health Record Data From the Medical Monitoring Device for Actual Monitoring at the Bedside in Bronchiolitis.
Description: This measure will be calculated using chart review (to determine presence of electronic health record data from the medical monitoring device) and direct observation (to determine actual monitoring at the bedside). This outcome compared EHR data at minute 0 (same minute as direct observation occurred). The numerator is the number of patients who were continuously monitored at the bedside.
  The denominator is the number of patients who had EHR data suggesting that they were continuously monitored.
Time Frame: 4 months
Population: The denominator for PPV calculation was the total number of patients who had EHR data suggesting that they were continuously monitored, which was 104 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | PATIENTS OBSERVED - Intervention (Single Arm)
Number analyzed (Participants) | 104
Participants | 92

8. Secondary Outcome: Negative Predictive Value of the Absence of Electronic Health Record Data From the Medical Monitoring Device for Absence of Monitoring at the Bedside in Bronchiolitis.
Description: This measure will be calculated using chart review (to determine presence of electronic health record data from the medical monitoring device) and direct observation (to determine actual monitoring at the bedside). This outcome compared EHR data at minute 0 (same minute as direct observation occurred). The numerator is the number of patients who were not observed to be continuously monitored at the bedside. The denominator is the number of patients who had EHR data suggesting that they were NOT continuously monitored.
Time Frame: 4 months
Population: The denominator for negative predictive value calculation was the total number of patients who had EHR data suggesting that they were NOT continuously monitored, which was 564 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | PATIENTS OBSERVED - Intervention (Single Arm)
Number analyzed (Participants) | 564
Participants | 554

ADVERSE EVENTS:
Time Frame: During 4-month active deimplementation study period.
Description: Systematic surveillance for PATIENTS:
  * Monitor for code blue /rapid response team activations in unmonitored bronchiolitis patients
  * Investigators determine whether the Adverse Event meets Serious Adverse Event (SAE)/unanticipated problem (UAP) criteria
  We did not conduct systematic assessment for Serious Adverse Events, Other (Not Including Serious) Adverse Events, code blue events, rapid response events, or all-cause mortality in STAFF SURVEYED.
Arm/Group | PATIENTS OBSERVED - Intervention (Single Arm) | STAFF SURVEYED - Intervention (Single Arm)
All-Cause Mortality (participants affected / at risk) | 0/1051 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1051 | 0/0
Other Adverse Events (participants affected / at risk) | 5/1051 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PATIENTS OBSERVED - Intervention (Single Arm) (N=1051) | STAFF SURVEYED - Intervention (Single Arm) (N=0)
a code blue or rapid response team activation - unmonitored patient (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) — a code blue or rapid response team call to a study unit for bronchiolitis in an unmonitored patient, determined not to be related to trial interventions. This AE does NOT apply to STAFF surveyed. Zero STAFF are at risk of this event.
a code blue or rapid response team activation - monitored patient (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — a code blue or rapid response team call to a study unit for bronchiolitis in a monitored patient, determined not to be related to trial interventions. This AE does NOT apply to STAFF surveyed. Zero STAFF are at risk of this event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT04178941/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT04178941/ICF_001.pdf